CLINICAL TRIAL: NCT06067906
Title: Weight Loss Following an Episode of Pre-eclampsia Using a Dissociated or Hypocaloric Diet in Overweight or Obese Patients
Acronym: POPADIPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHM-2022/S08/12
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pre-Eclampsia; Obesity
Keywords: pre-eclampsia; obesity; dissociated diet
MeSH Terms: conditions — Pre-Eclampsia; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator)
  Interventions: Other: Hypocaloric diet
- innovative group (Experimental)
  Interventions: Other: Dissociated diet

INTERVENTIONS:
Other: Hypocaloric diet — Hypocaloric diet
  Arms: control group
Other: Dissociated diet — Dissociated diet
  Arms: innovative group

SUMMARY:
In view of the known link between pre-eclampsia, overweight/obesity and chronic kidney disease, the aim is to offer for obese and overweight patients to reduce their BMI without reducing lean body mass.

The POPADIPE project will make it possible to limit overweight or obesity by means of nutritional management chosen by the patient (hypocaloric or a dissociated diet). The latter has been the subject of little scientific investigation, particularly in relation to the management of post-pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Person affiliated to social security
* Free, informed and written consent signed by the participant and the investigator (no later than the day of day of inclusion and before any examination required by the research)
* Patient over 18 years of age at the time of inclusion and < 45 years of age
* Having had an pre-eclampsia in the last 5 years according to the definitions of the ISSHP 2018
* Patient with a BMI between 25 kg/m² and 40 kg/m² who accepts dietetic follow up
* Patient with a medical prescription for dietetic follow-up aimed at losing weight loss
* Patient with a balanced diet

Exclusion Criteria:

* Patients with a mental disability or language barrier that prevents them from understanding or consenting to the study
* Patients deprived of their liberty by judicial or administrative decision
* Patients under psychiatric care
* Patients subject to a legal protection measure
* Patients with cognitive disorders or defined eating disorders
* Patients who are pregnant or breast-feeding
* Patients undergoing steroid treatment and/or immunosuppression
* Have been on a low-calorie or dissociated diet for at least 6 months
* Patients with CKD stage ≥ 3A

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2028-11-02 (Estimated); Study Completion 2028-11-02 (Estimated)

PRIMARY OUTCOMES:
Demonstrate Efficiency of personalised dietary management on weight loss in patients with a history of pre-eclampsia | 1 year after care
  Efficiency is evaluated by weight measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No